CLINICAL TRIAL: NCT03566264
Title: Characterizing the Acute Decompensated Heart Failure (ADHF) Patient Population in the United States (US)
Brief Title: Study of the Sudden Heart Failure Participant Population in the US
Status: Withdrawn | Type: Observational
Why Stopped: Program has been terminated.
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV013-031
Record Dates: First submitted 2018-04-24; First posted 2018-06-25 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Heart Decompensation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants hospitalized with ADHF
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
An observational study using data from a large US electronic health record database to find participants hospitalized with ADHF who do not have a concurring heart attack

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older on the index date
* At least 6 months of activity in the database
* An inpatient visit with at least one of the following ICD-9 or ICD-10 diagnosis codes (ICD-9 diagnosis codes: 428.xx, 785.51 or ICD-10 diagnosis codes: I50.xx, R57.0) in the primary or secondary position OR mention of "heart failure" on the admission record

Exclusion Criteria:

* An average LVEF ≥ 40 during the hospitalization
* Any code for myocardial infarction (ICD-9 diagnosis code: 410.xx, ICD-10 diagnosis code: I21.xx) or related terms such as "myocardial infarction", "mi", "infarct" or "heart attack" occurring during the index hospitalization

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be participants hospitalized with ADHF who do not have a coincident myocardial infarction and who have at least 6 months of activity in the database prior to the hospitalization
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Incidence of comorbid events among hospitalized ADHF participants | In the 30 days after discharge
Incidence of participants hospitalized with ADHF | Up to 66 months
Incidence of participants hospitalized with ADHF | In the 30 days after discharge
Incidence of comorbid events among hospitalized ADHF participants | Up to 66 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Bristol-Myers Squibb, Princeton, New Jersey
  - Local Institution, Princeton, New Jersey

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm